CLINICAL TRIAL: NCT03616730
Title: Validation of a Non-invasive Cardiac Output Monitor (NICOM) in Pregnant Women With Structural Heart Disease
Brief Title: NICOM in Pregnant Women With Heart Disease
Status: Terminated | Type: Observational
Why Stopped: PI leaving institution
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 18-062
Record Dates: First submitted 2018-07-25; First posted 2018-08-06 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Heart Diseases in Pregnancy; Congenital Heart Disease in Pregnancy
Keywords: Non-invasive cardiac output monitor; Cardiac output

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Heart Disease in pregnancy group: Fifty women will be recruited with structurally and functionally abnormal hearts without a history of chronic hypertension, pre-gestational diabetes, multiple gestations, preeclampsia, autoimmune disease, and anyone with a history of cardiomyopathy but currently normal ejection fraction. Women who are unable to give informed consent will not be included.
  Interventions: Diagnostic Test: NICOM (non-invasive cardiac output monitor)
- Control Group: Fifty women will be recruited with structurally normal hearts without a history of chronic hypertension, pre-gestational diabetes, multiple gestations, preeclampsia, autoimmune disease, and anyone with a history of cardiomyopathy but currently normal ejection fraction. Any woman on cardiac or antihypertensive medications (beta blockers, calcium channel blockers, hydralazine) will be excluded. Women who are unable to give informed consent will not be included.
  Interventions: Diagnostic Test: NICOM (non-invasive cardiac output monitor)

INTERVENTIONS:
Diagnostic Test: NICOM (non-invasive cardiac output monitor) — Transthoracic bio-reactance, or the non-invasive cardiac output measurement [NICOMTM, Cheetah Medical Inc., Portland, OR] system, is a new technique that is able to measure multiple hemodynamic parameters with four transdermal electrodes placed on the patients' thorax. It is based on frequency- and phase-modulation of the voltage signal measured in response to an applied transthoracic current. It has shown acceptable accuracy, precision and responsiveness for cardiac output monitoring in patients experiencing a wide-range of hemodynamic situations and is a FDA-approved device.

SUMMARY:
An accepted "gold standard" for hemodynamic monitoring in women with both healthy and diseased hearts is not currently available. Pregnancy is associated with significant hemodynamic changes, both during and following delivery, which can be even more profound in the structurally-abnormal heart. Clinical management of these women is based on surrogate markers of cardiac indices such as peripheral blood pressure, heart rate and oxygen saturation, rather than the use of invasive testing due to its associated complications. Echocardiography has largely replaced PAC in the obstetric population to measure cardiac output due to its non-invasive nature and good correlation with PAC18. However, its use is limited in the intrapartum period due to the need for clinical expertise in obtaining and interpreting the images. The proposed study has the potential to validate bio-reactance cardiac output monitoring using the NICOM against echocardiography for use in structurally normal and abnormal pregnant hearts in order to better drive goal-directed (specifically delivery mode) therapy through continuous hemodynamic monitoring during the second and third stages of labor, and 24 hours postpartum.

DETAILED DESCRIPTION:
Major hormonal and hemodynamic changes occur in the cardiovascular system in pregnancy that can unmask and impact underlying cardiac disease. Cardiac output can rise by up to 50% throughout gestation, with an additional 30% rise intrapartum. This increase is multifactorial, owing to an increase of 50% in maternal blood volume during pregnancy, a decrease in afterload due to a decline in systemic vascular resistance and a rise in the maternal heart rate of up to 20 beats per minute. Cardiac output has been the most extensively studied physiologic parameter of cardiac performance during pregnancy, and is dependent on both heart rate and stroke volume. Most of the changes in cardiac output on pregnancy are a result of stroke volume. However, during the mid-second trimester, stroke volume plateaus while heart rate continues to rise, becoming the major contributor to cardiac output in the latter half of pregnancy. During labor, cardiac output is further increased by the autotransfusion of blood from the uterus during a uterine contraction and maternal expulsive efforts. This can lead to an increase of up to 500cc of blood within seconds into the systemic circulation, which can significantly impact cardiac output and stroke volume.

Following delivery, many of these cardiovascular changes reverse in the first 2 weeks postpartum with further normalization toward preconception values 3-12 months later. Women without heart disease adapt well and adverse events are generally rare. However, the stress induced by these antenatal changes can cause a patient with underlying disease to decompensate during the latter half of pregnancy and more specifically, intrapartum when these changes peak. Studies on maternal morbidity attributable to cardiac disease in the United States have shown the most likely time for an adverse cardiac event is intrapartum and immediately postpartum, owing to the drastic and acute changes in hemodynamic status during these time periods. Without an invasive monitor (PAC), hemodynamic monitoring during these time relies on surrogate markers such as blood pressure or heart rate.

There is relatively scarce data on continuous hemodynamic profiles in women with both congenital and acquired heart disease in pregnancy, specifically during labor. Previous literature on the use of invasive monitoring (PAC) during pregnancy have been performed only intermittently during the labor and postpartum process. However, the hemodynamic status during the second and third labor stages is not static and therefore the need for continuous evaluation cannot be underscored.

The increased morbidity associated with invasive monitoring limits the use of pulmonary artery catheters in the pregnant population and therefore a non-invasive way to obtain hemodynamic profiles in women with heart disease is desirable. The non-invasive cardiac output monitor (NICOM) is based on bio-reactance technology and is operator-independent, allowing negligible inter-observer variability in data collection and ease of use. Measurements of cardiac output and stroke volume are not dependent on the distance between the electrodes, which can significantly increase the accuracy of the results. It involves the application of four sensors on the thorax. Changes in aortic blood flow drive phase shifts of propagating waves which are detected by the sensors as the frequency changes. These changes correlate with instantaneous changes in blood volume and blood flow in the aorta. Bio-reactance has been validated against pulmonary artery catheters in non-pregnant populations which manifest various forms of hemodynamic instability and following cardiac surgery.

Transthoracic bio-reactance, or the non-invasive cardiac output measurement [NICOMTM, Cheetah Medical Inc., Portland, OR] system, is a new technique that is able to measure multiple hemodynamic parameters with four transdermal electrodes placed on the patients' thorax. It is based on frequency- and phase-modulation of the voltage signal measured in response to an applied transthoracic current. Its readings have been shown in multiple studies to correlate well with PAC in the non-pregnant population. It has shown acceptable accuracy, precision and responsiveness for cardiac output monitoring in patients experiencing a wide-range of hemodynamic situations. However, it has not been validated in the pregnant, structurally abnormal heart i.e. congenital cardiac disease, as this was exclusion criteria in the aforementioned studies. Establishing normative values during the second stage of labor utilizing the NICOM in women with congenital cardiac disease has the potential to be clinically useful in developing goal-directed management therapy for these women.

ELIGIBILITY:
Inclusion Criteria:

* CONTROL GROUP:
* singleton pregnancy
* > 18 years of age
* enrolled in first trimester of pregnancy
* planning delivery at Saint Luke's Hospital of Kansas City
* STUDY GROUP:
* history of either congenital or acquired heart disease
* singleton pregnancy
* > 18 years of age
* enrolled in first trimester of pregnancy
* planning delivery at Saint Luke's Hospital of Kansas City

Exclusion Criteria:

Control group:

* no history of either acquired or congenital heart disease
* no hypertension, diabetes, multiple gestations, preeclampsia, or autoimmune disease
* no use of antihypertensive medications
* inability to give informed consent

Study Group:

* no hypertension, diabetes, multiple gestations, preeclampsia, autoimmune disease
* inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women.
Study Population: Both healthy pregnant women and pregnant women with a history of heart disease will be recruited to participate in our observational, non-inferiority trial comparing the cardiac output measurements obtained by two different modalities. Women in their first trimester will be approached to participate. Any woman with a history of either structural or acquired heart disease will be recruited into the study group as described above. Women with structurally normal hearts in the first trimester who meet the aforementioned inclusion criteria will also be recruited to participate as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Non-inferiority between NICOM and echocardiogram cardiac output measurements | 3 year recruitment
  We will compare the cardiac output measurements obtained from the NICOM in each trimester with those obtained from the echocardiogram. We expect a mean percentage difference of < 30% between modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Florio, DO, Principal Investigator — Saint Luke's Hospital of Kansas City/UMKC Assistant Professor, MFM Division
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Canobbio MM, Warnes CA, Aboulhosn J, Connolly HM, Khanna A, Koos BJ, Mital S, Rose C, Silversides C, Stout K; American Heart Association Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; Council on Functional Genomics and Translational Biology; and Council on Quality of Care and Outcomes Research. Management of Pregnancy in Patients With Complex Congenital Heart Disease: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2017 Feb 21;135(8):e50-e87. doi: 10.1161/CIR.0000000000000458. Epub 2017 Jan 12. PMID 28082385
- [Background] Velissaris D, Karamouzos V, Kotroni I, Pierrakos C, Karanikolas M. The Use of Pulmonary Artery Catheter in Sepsis Patients: A Literature Review. J Clin Med Res. 2016 Nov;8(11):769-776. doi: 10.14740/jocmr2719w. Epub 2016 Sep 29. PMID 27738477
- [Background] Cornette J, Laker S, Jeffery B, Lombaard H, Alberts A, Rizopoulos D, Roos-Hesselink JW, Pattinson RC. Validation of maternal cardiac output assessed by transthoracic echocardiography against pulmonary artery catheterization in severely ill pregnant women: prospective comparative study and systematic review. Ultrasound Obstet Gynecol. 2017 Jan;49(1):25-31. doi: 10.1002/uog.16015. Epub 2016 Nov 28. PMID 27404397
- [Background] Ohashi Y, Ibrahim H, Furtado L, Kingdom J, Carvalho JC. Non-invasive hemodynamic assessment of non-pregnant, healthy pregnant and preeclamptic women using bioreactance. [corrected]. Rev Bras Anestesiol. 2010 Nov-Dec;60(6):603-13, 335-40. doi: 10.1016/S0034-7094(10)70075-1. English, Portuguese, Spanish. PMID 21146056
- [Background] Keren H, Burkhoff D, Squara P. Evaluation of a noninvasive continuous cardiac output monitoring system based on thoracic bioreactance. Am J Physiol Heart Circ Physiol. 2007 Jul;293(1):H583-9. doi: 10.1152/ajpheart.00195.2007. Epub 2007 Mar 23. PMID 17384132
- [Background] Squara P, Denjean D, Estagnasie P, Brusset A, Dib JC, Dubois C. Noninvasive cardiac output monitoring (NICOM): a clinical validation. Intensive Care Med. 2007 Jul;33(7):1191-1194. doi: 10.1007/s00134-007-0640-0. Epub 2007 Apr 26. PMID 17458538
- [Background] Vinayagam D, Patey O, Thilaganathan B, Khalil A. Cardiac output assessment in pregnancy: comparison of two automated monitors with echocardiography. Ultrasound Obstet Gynecol. 2017 Jan;49(1):32-38. doi: 10.1002/uog.15915. PMID 26970353
- [Background] McLaughlin K, Wright SP, Kingdom JCP, Parker JD. Clinical Validation of Non-Invasive Cardiac Output Monitoring in Healthy Pregnant Women. J Obstet Gynaecol Can. 2017 Nov;39(11):1008-1014. doi: 10.1016/j.jogc.2017.02.015. Epub 2017 Jul 18. PMID 28733057
- [Background] Roberts LA, Ling HZ, Poon LC, Nicolaides KH, Kametas NA. Maternal hemodynamics, fetal biometry and Doppler indices in pregnancies followed up for suspected fetal growth restriction. Ultrasound Obstet Gynecol. 2018 Oct;52(4):507-514. doi: 10.1002/uog.19067. PMID 29607557
- [Background] Sandham JD, Hull RD, Brant RF, Knox L, Pineo GF, Doig CJ, Laporta DP, Viner S, Passerini L, Devitt H, Kirby A, Jacka M; Canadian Critical Care Clinical Trials Group. A randomized, controlled trial of the use of pulmonary-artery catheters in high-risk surgical patients. N Engl J Med. 2003 Jan 2;348(1):5-14. doi: 10.1056/NEJMoa021108. PMID 12510037
- [Background] Mabie WC, DiSessa TG, Crocker LG, Sibai BM, Arheart KL. A longitudinal study of cardiac output in normal human pregnancy. Am J Obstet Gynecol. 1994 Mar;170(3):849-56. doi: 10.1016/s0002-9378(94)70297-7. PMID 8141215
- [Background] Hunter S, Robson SC. Adaptation of the maternal heart in pregnancy. Br Heart J. 1992 Dec;68(6):540-3. doi: 10.1136/hrt.68.12.540. PMID 1467047
- [Background] Dyer RA, James MF. Maternal hemodynamic monitoring in obstetric anesthesia. Anesthesiology. 2008 Nov;109(5):765-7. doi: 10.1097/ALN.0b013e31818a3825. No abstract available. PMID 18946283
- [Background] Engoren M, Barbee D. Comparison of cardiac output determined by bioimpedance, thermodilution, and the Fick method. Am J Crit Care. 2005 Jan;14(1):40-5. PMID 15608107
- [Background] Lee W, Rokey R, Cotton DB. Noninvasive maternal stroke volume and cardiac output determinations by pulsed Doppler echocardiography. Am J Obstet Gynecol. 1988 Mar;158(3 Pt 1):505-10. doi: 10.1016/0002-9378(88)90014-2. PMID 3348311
- [Background] Easterling TR, Watts DH, Schmucker BC, Benedetti TJ. Measurement of cardiac output during pregnancy: validation of Doppler technique and clinical observations in preeclampsia. Obstet Gynecol. 1987 Jun;69(6):845-50. PMID 3574814
- [Background] Critchley LA, Critchley JA. A meta-analysis of studies using bias and precision statistics to compare cardiac output measurement techniques. J Clin Monit Comput. 1999 Feb;15(2):85-91. doi: 10.1023/a:1009982611386. PMID 12578081
- [Background] Doherty A, El-Khuffash A, Monteith C, McSweeney L, Breatnach C, Kent E, Tully E, Malone F, Thornton P. Comparison of bioreactance and echocardiographic non-invasive cardiac output monitoring and myocardial function assessment in primagravida women. Br J Anaesth. 2017 Apr 1;118(4):527-532. doi: 10.1093/bja/aex045. PMID 28403411
- [Background] Vinayagam D, Bowe S, Sheehan E, Thilaganathan B, Khalil A. Non-Invasive Haemodynamic Monitoring in Pregnancy: A Comparative Study Using Ultrasound and Bioreactance. Fetal Diagn Ther. 2017;41(4):273-282. doi: 10.1159/000446650. Epub 2016 Oct 6. PMID 27705969
- See also: Up to Date article — http://uptodate.com/contents/acquired-heart-disease-and-pregnancy?topicKey=Cardiology